CLINICAL TRIAL: NCT05003882
Title: A Randomized, Open-label Study of Commercially Available, Orally Ingestible, Cannabidiol (CBD) Products Used in the Real-world Setting for Pain, Sleep, and Anxiety
Brief Title: Radicle ACES: A Study of Commercially Available CBD Used in the Real-world Setting
Acronym: RWE-ACES
Status: Completed | Type: Observational
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Other Study IDs: Radicle; RADX-2021-002 (Other: Radicle)
Record Dates: First submitted 2021-07-23; First posted 2021-08-13 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Pain; Sleep Disturbance; Anxiety
MeSH Terms: conditions — Pain; Parasomnias; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (14):
- Arm A: Commercially available, orally ingestible CBD product A
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm B: Commercially available, orally ingestible CBD product B
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm C: Commercially available, orally ingestible CBD product C
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm D: Commercially available, orally ingestible CBD product D
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm E: Commercially available, orally ingestible CBD product E
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm F: Commercially available, orally ingestible CBD product F
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm G: Commercially available, orally ingestible CBD product G
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm H: Commercially available, orally ingestible CBD product H
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm I: Commercially available, orally ingestible CBD product I
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm J: Commercially available, orally ingestible CBD product J
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm K: Commercially available, orally ingestible CBD product K
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm L: Commercially available, orally ingestible CBD product L
  Interventions: Other: Commercially available, orally ingestible CBD product
- Arm M: Commercially available, orally ingestible CBD product M
  Interventions: Other: Commercially available, orally ingestible CBD product
- Control: Waitlist control

INTERVENTIONS:
Other: Commercially available, orally ingestible CBD product — botanically-derived CBD extract product
  Groups: Arm A; Arm B; Arm C; Arm D; Arm E; Arm F; Arm G; Arm H; Arm I; Arm J; Arm K; Arm L; Arm M

SUMMARY:
A randomized, open-label study of commercially available, orally ingestible, Cannabidiol (CBD) products used in the real-world setting for pain, sleep, and anxiety.

DETAILED DESCRIPTION:
Radicle ACES is a real-world evidence study that aims to determine the effect of CBD on overall well-being, anxiety, sleep, and pain over a 28-day period in treatment groups compared to a waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 21 years of age
* Live in the USA
* Endorse symptoms of anxiety, chronic pain, or sleep disturbances as a primary reason for taking a CBD product
* Must have regular access to a computer, mobile device, and/or the internet to complete surveys

Exclusion Criteria:

* A person pregnant, trying to become pregnant or breastfeeding
* Anyone diagnosed with liver disease or considered a heavy drinker
* Anyone taking medication that warns against grapefruit consumption

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (21 yo and older) living in the USA
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Greater increase in overall well-being from baseline | 4 weeks
  Overall well-being as assessed by KEMP Quality of Life Scale (QOL scale 1-7 where 7 is a better QOL)
Improvement in overall well-being from baseline | 4 weeks
  Overall well-being as assessed by World Health Organization (WHO) 5 Well Being Index (0-5 where 5 is better well-being)
Change in overall well-being from baseline | 4 weeks
  Overall well-being as assessed by Patient Global Impression of Change (PGIC statement selection much improved to much worse)

SECONDARY OUTCOMES:
Improvement in sleep from baseline | 4 weeks
  Sleep as assessed by PROMIS (Patient Reported Outcome Measurement Information System) Sleep Short Form 8B (scale 1-5 where a 5 represents worse sleep)
Change in sleep from baseline | 4 weeks
  Sleep as assessed by PGIC (statement selection much improved to much worse)
Change in anxiety from baseline | 4 weeks
  Anxiety as assessed by PGIC (statement selection much improved to much worse)
Less anxiety from baseline | 4 weeks
  Anxiety as assessed by GAD-7 (scale 0-3 where 3 is greater anxiety)
Decrease in anxiety from baseline | 4 weeks
  Anxiety as assessed by PROMIS Anxiety 4A (scale 1-5 where 5 is greater anxiety)
Less pain relative to baseline | 4 weeks
  Pain as assessed by PEG (scale 1-10 where a higher score is greater pain)
Change in pain from baseline | 4 weeks
  Pain as assessed by PGIC (statement selection much improved to much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Laird, PhD, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science, Encinitas, California, United States

IPD SHARING:
Plan to Share IPD: No
only aggregated and anonymized data will be shared.